CLINICAL TRIAL: NCT04641299
Title: A Randomized, Parallel, Double-blind, Placebo-controlled, Dose-ranging, Phase 2b Study to Evaluate the Efficacy, Safety and Tolerability of AZD8233 Treatment in Participants With Dyslipidemia
Brief Title: A Study of AZD8233 in Participants With Dyslipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7990C00003
Record Dates: First submitted 2020-10-28; First posted 2020-11-23 (Actual); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Dyslipidaemia
Keywords: Dose Range Finding; AZD8233; Efficacy; PK; PD; Immunogenicity; Safety; Tolerability
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo solution for subcutaneous injection.
  Interventions: Drug: Placebo
- AZD8233 high dose (Experimental): AZD8233 high dose for subcutaneous injection.
  Interventions: Drug: AZD8233
- AZD8233 medium dose (Experimental): AZD8233 medium dose for subcutaneous injection.
  Interventions: Drug: AZD8233
- AZD8233 low dose (Experimental): AZD8233 low does for subcutaneous injection.
  Interventions: Drug: AZD8233

INTERVENTIONS:
Drug: AZD8233 — PCSK9-targeted ASO for the reduction of circulating levels of LDL-C.
  Arms: AZD8233 high dose; AZD8233 low dose; AZD8233 medium dose
Drug: Placebo — Placebo solution
  Arms: Placebo

SUMMARY:
AZD8233 is a PCSK9-targeted ASO for the reduction of circulating levels of LDL-C. This study aims to evaluate the dose-dependent reduction in LDL-C after SC administration of multiple doses of AZD8233 as well as the associated adverse effects profile. The data generated will be used to guide choice of doses, dosing regimens, and sample sizes, as well as safety and PD monitoring in the further clinical development program.

DETAILED DESCRIPTION:
This is a randomized parallel, double-blind, placebo-controlled, dose-ranging Phase 2b study in approximately 108 participants with dyslipidemia. The primary objective of the study is to investigate the effect of AZD8233 on LDL-C across different dose levels. The study will be conducted at up to 25 sites in up to 4 countries.

The screening period starts up to 42 days before the randomization visit and ends on Day -1. Eligible participants will attend 7 visits during the treatment period and 7 additional visits during the safety follow up period. Eligible participants are randomized across four different treatment arms in a 1:1:1:1 ratio for a 12-week treatment period. The planned treatment arms are AZD8233 low dose, AZD8233 medium dose, AZD8233 high dose, and Placebo. Participants will be dosed SC on Days 1, 8, 29, and 57.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female.
* Participant must be 18 to 75 years of age.
* Body mass index between 19 and 40 kg/m2.
* Participants who have a fasting LDL-C ≥ 70 mg/dL but < 190 mg/dL.
* Have fasting triglycerides < 400 mg/dL.
* Should be receiving moderate- or high-intensity statin therapy.
* Should be on stable medication for ≥ 3 months prior to screening with no planned medication or dose change during study participation. The exception to this restriction is for fenofibrate; if the participant is receiving fenofibrate, the therapy must be stable for at least 6 weeks prior to randomization at a dose that is appropriate for the duration of the study in the judgement of the Investigator. Other fibrate therapy (and derivatives) are prohibited.

Key Exclusion Criteria:

* Estimated glomerular filtration rate < 40 mL/min/1.73m2 CKD-EPI.
* Any uncontrolled or serious disease, or any medical dysfunction or surgical condition that, in the opinion of the Investigator, may either interfere with participation in the clinical study and/or put the participant at significant risk.
* Poorly controlled type 2 diabetes mellitus, defined as HbA1c > 10% at Visit 1.
* Acute ischaemic cardiovascular event in the last 12 months prior to randomization.
* Heart failure with New York Heart Association (NYHA) Class III-IV.
* High-risk of bleeding as judged by the Investigator.
* Malignancy (except non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal
* Carcinoma in-situ, or Stage 1 prostate carcinoma) within the last 10 years.
* LDL or plasma apheresis within 12 months prior to randomization.
* Uncontrolled hypertension defined as average supine SBP > 160 mmHg or DBP > 90 mmHg at Visit 1 or Visit 3.
* Heart rate after 10 minutes supine rest < 50 bpm or > 100 bpm.
* Any laboratory values with the following deviations at Screening:

  * Positive result on screening for hepatitis B, hepatitis C or HIV.
  * ALT > 1.5 × ULN.
  * AST > 1.5 × ULN.
  * TBL > ULN.
  * ALP > 1.5 × ULN.
  * WBC < LLN.
  * Haemoglobin < 12 g/dL in men or < 11 g/dL in women.
  * Platelet count ≤ LLN.
  * aPTT > ULN and PT > ULN.
  * UACR > 11.3 mg/mmol (100 mg/g).
  * UPCR > 300 mg/g.
* Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities in the 12-lead ECG as judged by the Investigator.
* Mipomersen, or lomitapide within 12 months prior to randomization.
* Previous administration of AZD8233/AZD6615.
* Previous administration of PCSK9 inhibition treatment.
* Participation in another clinical study with a study intervention administered in the last 3 months prior to randomization or 5 half-lives from last dose to first administration of study intervention, whichever is the longest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (10):
  - Research Site, Roseville, California
  - Research Site, Inverness, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Meridian, Idaho
  - Research Site, Indianapolis, Indiana
  - Research Site, New Windsor, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
- Denmark (5):
  - Research Site, Aarhus N
  - Research Site, Frederiksberg
  - Research Site, Herlev
  - Research Site, Roskilde
  - Research Site, Viborg
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Rožňava
  - Research Site, Trebišov

REFERENCES:
- [Derived] Clewe O, Rekic D, Quartino AL, Carlsson B, Higashimori M, Wernevik L, Hofherr A, Ryden-Bergsten T, Nilsson C, Knochel J. Population pharmacokinetics of a novel PCSK9 antisense oligonucleotide. Br J Clin Pharmacol. 2024 Jun;90(6):1503-1513. doi: 10.1111/bcp.16046. Epub 2024 Mar 19. PMID 38504437
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00003&attachmentIdentifier=1cdc0745-522a-48f6-8af1-2c8331bc5ac2&fileName=d7990c00003_CSP_Redacted.pdf&versionIdentifier=
- See also: redacted Statistical Analysis Plan — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00003&attachmentIdentifier=5e58110c-0521-493c-85d4-8fff83651138&fileName=D7990C00003_SAP_Redacted.pdf&versionIdentifier=
- See also: Redacted Clinical Study Report Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7990C00003&attachmentIdentifier=e0de9a3b-3e99-46dd-a46f-c217b8279d7e&fileName=d7990c00003_CSR_synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 19 clinical research center in Denmark, Slovakia and the USA. First subject enrolled (First subject first visit/first consent signed date): 28 October 2020. Last subject last visit: 20 July 2021.
Groups:
- AZD8233 Low Dose: AZD8233 low dose for subcutaneous injection.
Period: Overall Study
Arm/Group | AZD8233 Low Dose | AZD8233 Medium Dose | AZD8233 High Dose | Placebo
Started | 30 | 30 | 29 | 30
Completed | 28 | 29 | 27 | 30
Not Completed | 2 | 1 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Reason not given | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose | Placebo | Total
Number analyzed (Participants) | 29 | 30 | 30 | 30 | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.4 (8.4) | 60.6 (7.4) | 61.8 (7.1) | 63.9 (7.3) | 61.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 16 | 18 | 57
  Male | 18 | 18 | 14 | 12 | 62
Race/Ethnicity, Customized [Number; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 0
  ASIAN | 0 | 0 | 1 | 0 | 1
  BLACK OR AFRICAN AMERICAN | 1 | 2 | 2 | 3 | 8
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0 | 0 | 0
  WHITE | 28 | 28 | 27 | 27 | 110

OUTCOME MEASURES:

1. Primary Outcome: Change in Low-density Lipoprotein Cholesterol (LDL-C) at Week 12.
Description: Change from baseline in low-density lipoprotein cholesterol (LDL-C) at week 12. Results are based on Mixed Model Repeated Measures (MMRM) analysis on the log-transformed change from baseline. Log-transformed change from baseline is calculated as the visit value in log minus the baseline value in log. The results from the model are then back transformed.
Time Frame: Baseline to week 12
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 26 | 26 | 28 | 27
Ratio | 0.978 [0.834 to 1.147] | 0.206 [0.174 to 0.242] | 0.270 [0.230 to 0.317] | 0.606 [0.517 to 0.710]

2. Secondary Outcome: Relative Change From Baseline in PCSK9 Concentration in Plasma at Week 12.
Description: Relative change from baseline in PCSK9 concentration in plasma at week 12.
Time Frame: Baseline to week 12
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 27 | 26 | 28 | 28
Ratio | 0.950 [0.770 to 1.180] | 0.060 [0.050 to 0.080] | 0.110 [0.090 to 0.140] | 0.420 [0.340 to 0.520]

3. Secondary Outcome: Percentage Change From Baseline in Concentration of TC, HDL-C, Non-HDL-C, VLDL-C, ApoA1, ApoB, Lp(a), Triglycerides, Remnants Cholesterol
Description: Percentage change from baseline in concentration of TC, HDL-C, Non-HDL-C, VLDL-C, ApoA1, ApoB, Lp(a), Triglycerides, Remnants cholesterol at week 12
Time Frame: Baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 26 | 26 | 28 | 28
Percent
  Triglycerides | 2.69 [-8.19 to 13.56] | -12.70 [-23.88 to -1.52] | -12.95 [-23.77 to -2.12] | -7.70 [-18.44 to 3.05]
  Total cholesterol | -1.11 [-6.56 to 4.35] | -47.58 [-53.37 to -41.78] | -43.90 [-49.43 to -38.37] | -21.13 [-26.56 to -15.70]
  HDL-C | 1.34 [-3.28 to 5.97] | 5.57 [0.90 to 10.25] | 6.50 [1.96 to 11.04] | 3.37 [-1.12 to 7.86]
  Non-HDL-C | -0.65 [-7.81 to 6.51] | -67.92 [-75.38 to -60.45] | -61.25 [-68.38 to -54.11] | -29.57 [-36.58 to -22.56]
  VLDL-C | 3.22 [-7.90 to 14.35] | -11.13 [-22.59 to 0.33] | -12.09 [-23.04 to -1.15] | -7.54 [-18.36 to 3.27]
  ApoB | -1.65 [-7.83 to 4.53] | -67.07 [-73.46 to -60.68] | -60.13 [-66.33 to -53.93] | -29.50 [-35.64 to -23.35]
  Lp(a) | 31.22 [-2.88 to 65.33] | -37.74 [-72.02 to -3.46] | -36.64 [-70.69 to -2.59] | -6.02 [-40.62 to 28.58]
  Remnants cholesterol | 6.38 [-20.28 to 33.05] | -26.84 [-54.23 to 0.54] | -16.54 [-42.97 to 9.88] | -13.50 [-39.57 to 12.56]

4. Secondary Outcome: Plasma Concentration of AZD8233
Description: Plasma concentration of AZD8233 after first dose administration
Time Frame: Measurement at week 1, week 4, week 6, week 8, week 10, week 12, week 16, week 20, week 24 after first dose administration.
Population: No analysis made for placebo group.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 29 | 30 | 30
ug/L
  Week 1: number analyzed (Participants) | 25 | 28 | 28
  Week 1 | 1.201 (0.49) | 0.681 (0.24) | 0.346 (0.59)
  Week 4: number analyzed (Participants) | 24 | 27 | 29
  Week 4 | 1.366 (0.71) | 0.699 (0.33) | 0.238 (0.21)
  Week 6: number analyzed (Participants) | 25 | 27 | 30
  Week 6 | 1.917 (1.09) | 0.870 (0.34) | 0.288 (0.21)
  Week 8: number analyzed (Participants) | 24 | 27 | 28
  Week 8 | 1.000 (0.68) | 0.628 (0.57) | 0.152 (0.10)
  Week 10: number analyzed (Participants) | 25 | 27 | 30
  Week 10 | 1.562 (0.84) | 0.751 (0.29) | 0.241 (0.15)
  Week 12: number analyzed (Participants) | 26 | 28 | 28
  Week 12 | 0.976 (0.75) | 0.476 (0.23) | 0.134 (0.07)
  Week 16: number analyzed (Participants) | 26 | 27 | 29
  Week 16 | 0.507 (0.70) | 0.297 (0.53) | 0.087 (0.09)
  Week 20: number analyzed (Participants) | 24 | 28 | 28
  Week 20 | 0.376 (0.68) | 0.153 (0.26) | 0.053 (0.004)
  Week 24: number analyzed (Participants) | 24 | 27 | 29
  Week 24 | 0.350 (0.62) | 0.111 (0.15) | 0.111 (0.31)

5. Secondary Outcome: Anti-drug Antibodies (ADAs) During the Treatment Period and Follow-up Period
Description: ADA titre results for subjects with positive ADA during the treatment period and follow-up period.
Time Frame: Measurement at week 0, week 1, week 4, week 8, week 12, week 16, week 20, week 24
Population: Number Analyzed per Row reflects the study participants with positive ADA results at each time point.
Measure: Median (Full Range); unit: ADA titre
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 1 | 3 | 5 | 4
ADA titre
  Baseline: number analyzed (Participants) | 1 | 0 | 1 | 3
  Baseline | 100 [100 to 100] |  | 200 [200 to 200] | 100 [100 to 100]
  Week 1: number analyzed (Participants) | 1 | 0 | 1 | 4
  Week 1 | 100 [100 to 100] |  | 200 [200 to 200] | 100 [50 to 800]
  Week 4: number analyzed (Participants) | 1 | 2 | 3 | 4
  Week 4 | 100 [100 to 100] | 75 [50 to 100] | 200 [100 to 400] | 150 [100 to 1600]
  Week 8: number analyzed (Participants) | 1 | 2 | 3 | 3
  Week 8 | 100 [100 to 100] | 75 [50 to 100] | 200 [100 to 400] | 400 [200 to 3200]
  Week 12: number analyzed (Participants) | 1 | 2 | 4 | 3
  Week 12 | 50 [50 to 50] | 200 [200 to 200] | 200 [100 to 400] | 200 [200 to 1600]
  Week 16: number analyzed (Participants) | 1 | 2 | 4 | 3
  Week 16 | 100 [100 to 100] | 300 [200 to 400] | 200 [50 to 400] | 400 [100 to 1600]
  Week 20: number analyzed (Participants) | 1 | 2 | 5 | 3
  Week 20 | 100 [100 to 100] | 500 [200 to 800] | 200 [100 to 400] | 400 [200 to 1600]
  Week 24: number analyzed (Participants) | 1 | 3 | 4 | 3
  Week 24 | 100 [100 to 100] | 200 [50 to 800] | 300 [100 to 400] | 400 [200 to 800]

6. Secondary Outcome: Percentage Change From Baseline in Levels of LDL-C in Plasma
Description: Percentage change from baseline in levels of LDL-C in plasma from baseline to week 12.
Time Frame: Baseline to week 12
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 26 | 26 | 28 | 27
Percent | -1.53 [-9.14 to 6.09] | -76.50 [-84.37 to -68.63] | -69.26 [-76.89 to -61.63] | -32.22 [-39.79 to -24.66]

7. Other Pre Specified Outcome: Number of Subjects With an ECG Determined to be Abnormal and Clinically Significant
Description: Number of subjects with an ECG determined to be abnormal and clinically significant at baseline and end of treatment.
Time Frame: Baseline to Week 24
Measure: Number; unit: Number of subjects
Arm/Group | Placebo | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose
Number analyzed (Participants) | 30 | 29 | 30 | 30
Number of subjects
  Baseline | 0 | 0 | 0 | 0
  End of treatment | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of first IP dose throughout the treatment period of 12 weeks and including the follow-up period of 12 weeks - a total of 24 weeks. Serious AEs were recorded from the time of signature of informed consent.
Arm/Group | AZD8233 High Dose | AZD8233 Medium Dose | AZD8233 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/30 | 1/30 | 0/30
Other Adverse Events (participants affected / at risk) | 20/29 | 17/30 | 14/30 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8233 High Dose (N=29) | AZD8233 Medium Dose (N=30) | AZD8233 Low Dose (N=30) | Placebo (N=30)
Covid-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD8233 High Dose (N=29) | AZD8233 Medium Dose (N=30) | AZD8233 Low Dose (N=30) | Placebo (N=30)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asymptomatic covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal vestibulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipids increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/99/NCT04641299/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT04641299/SAP_001.pdf